CLINICAL TRIAL: NCT04599465
Title: A Phase 3b Open-label Study to Assess the Effect of Elexacaftor (ELX)/Tezacaftor (TEZ)/Ivacaftor (IVA) on Glucose Tolerance in Cystic Fibrosis Subjects With Abnormal Glucose Metabolism
Brief Title: A Study to Assess the Effect of ELX/TEZ/IVA on Glucose Tolerance in Participants With Cystic Fibrosis (CF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX19-445-117; 2020-003170-44 (EudraCT Number)
Record Dates: First submitted 2020-10-21; First posted 2020-10-22 (Actual); Results first posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ELX/TEZ/IVA (Experimental): Participants received ELX 200 mg /TEZ 100 mg /IVA 150 mg in the morning and IVA 150 mg in the evening.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed dose combination (FDC) tablets for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
Drug: IVA — Tablets for oral administration.
  Other Names: VX-770; ivacaftor

SUMMARY:
This study was evaluate the effect of elexacaftor (ELX)/tezacaftor (TEZ)/ivacaftor (IVA) on glucose tolerance in CF participants, 12 years of age and older who are heterozygous for the F508del mutation and a minimal function mutation (F/MF genotypes), with abnormal glucose metabolism.

ELIGIBILITY:
Key Inclusion Criteria:

* Heterozygous for F508del and an MF mutation (F/MF genotypes)
* Forced expiratory volume in 1 second (FEV1) value ≥ 30% of predicted mean for age, sex, and height
* Abnormal glucose tolerance determined by an OGTT as either:

  * Impaired glucose tolerance (IGT) defined as 2 hour post OGTT blood glucose level ≥140 to <200 mg/dL (≥7.77 to <11.10 mmol/L) and fasting blood glucose level <126 mg/dL (<7.00 mmol/L)
  * CF-related diabetes (CFRD) defined as either fasting hyperglycemia (blood glucose level ≥126 mg/dL [≥7.00 mmol/L] after an 8-hour fast) or 2-hour post OGTT blood glucose level ≥200 mg/dL (≥11.10 mmol/L)

Key Exclusion Criteria:

* Clinically significant liver cirrhosis with or without portal hypertension
* Solid organ or hematological transplantation
* Lung infection with organisms associated with a more rapid decline in pulmonary status
* Type 1 or Type 2 diabetes
* Duration of CFRD ≥5 years

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- Australia (9):
  - Royal Adelaide Hospital, Adelaide
  - The Prince Charles Hospital, Chermside
  - Alfred Hospital, Melbourne
  - Telethon Kids Institute, Nedlands
  - The Royal Children's Hospital, Parkville, VIC
  - Sydney Children's Hospital, Randwick
  - Mater Adult Hospital, South Brisbane
  - Queensland Children's Hospital, South Brisbane
  - Westmead Hospital, Westmead
- Belgium (3):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Czechia (2):
  - Klinika Nemoci Plicnich a Tuberkulozy, Brno
  - Fakultni nemocnice v Motole, Prague
- France (10):
  - Centre Hospitalier Intercommunal Creteil, Créteil
  - CHRU de Lille - Hopital Albert Calmette, Lille
  - CHU Marseille - Hopital Nord, Marseille
  - Hopital Arnaud de Villeneuve, Montpellier
  - Centre Hospitalier Universitaire De Nantes - G. R. Laennec, Nantes
  - Centre Hospitalier Universitaire (CHU) de Nice - Hopital Pasteur, Nice
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Rouen - Hopital Charles Nicolle, Rouen Cedex, Seine Maritime
  - Hopitaux Universitaires de Strasbourg, Strasbourg
  - Hopital Foch (Suresnes), Hopital Foch, Adultes, Suresnes
- Italy (6):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona
  - IRCCS Istituto Giannina Gaslini-Ospedale Pediatrico, Genova
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliero Universitaria Federico II Napoli, Naples
  - Azienda Ospedaliera di Verona - Ospedale Civile Maggiore, Verona
- Netherlands (4):
  - Academisch Medisch Centrum (Academic Medical Centre), Amsterdam
  - University Medical Center, Utrecht, Department of Pulmonology and Tuberculosis, Heidelberglaan
  - Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis van den Haag, The Hague
- Spain (7):
  - Hospital Saint Joan de Deu, Barcelona
  - Hospital Universitari Vall d Hebron, Barcelona
  - Hospital Universitari Vall d´Hebron Servicio de Broncoscopia, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

REFERENCES:
- [Derived] Durieu I, Clements B, Fabrizzi B, Mall MA, McKone E, Ramsey B, Tullis E, Taylor-Cousar JL, van der Meer R, Bachman E, Chin A, Conner S, Jennings M, Weinstock T, Colombo C, Robinson P. Impact of Elexacaftor/Tezacaftor/Ivacaftor on Glucose Tolerance and Abnormal Glucose Metabolism: A Phase 3b, Open-Label Clinical Trial. Am J Respir Crit Care Med. 2025 Oct;211(10):1926-1934. doi: 10.1164/rccm.202411-2312OC. PMID 40788823

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted in participants with cystic fibrosis (CF) aged 12 years and older who are heterozygous for the F508del mutation and a minimal function mutation (F/MF genotypes), with abnormal glucose metabolism.
Groups:
- ELX/TEZ/IVA: Participants received elexacaftor (ELX) 200 mg/tezacaftor (TEZ)100 mg ivacaftor (IVA) 150 mg in the morning and IVA 150 mg in the evening.
Period: Overall Study
Arm/Group | ELX/TEZ/IVA
Started | 69
Completed | 66
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal of consent (not due to AE) | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug during the treatment period were included in the baseline analysis.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 69
Age, Customized [Count of Participants; unit: Participants]
  Less than (<)18 years | 19
  More than or equal to (≥)18 years | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 41
  Not collected per local regulations | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 48
  Black or African American | 0
  Asian | 0
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 0
  Other | 1
  Not collected per local regulations | 20
2-hour Post-OGTT Blood Glucose Levels [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dl)] — Baseline 2-hour post-Oral Glucose Tolerance Test (OGTT) blood glucose level was defined as the average of valid pre-dose measurements at screening and Day 1. OGTT results were considered valid only when the participant was fasting for at least 8 hours.
  milligrams per deciliter (mg/dl) | 217.6 (73.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 2-hour Blood Glucose Levels Following an OGTT to the Average of Week 36 and Week 48
Description: Baseline 2-hour post-OGTT blood glucose level was defined as the average of valid pre-dose measurements at screening and Day 1. OGTT results were considered valid only when the participant was fasting for at least 8 hours.
Time Frame: Baseline, Week 36 and 48
Population: The Full Analysis Set (FAS) will include all enrolled participants who carry the intended CFTR allele mutation and have received at least 1 dose of study drug. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams per deciliter (mg/dl)
Groups:
- ELX/TEZ/IVA: Participants received ELX 200 mg /TEZ 100 mg/IVA 150 mg in the morning and IVA 150 mg in the evening.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 66
milligrams per deciliter (mg/dl) | -35.0 [-49.2 to -20.7]

2. Secondary Outcome: Percentage of Participants With Improvement in Dysglycemia Categorization at Week 48
Description: Baseline dysglycemia category was defined as the most recent non-missing measurement before the first dose of study drug in the treatment period. Improvement in dysglycemia is a change from cystic fibrosis-related diabetes (CFRD) at baseline to impaired glucose tolerance (IGT)/normal glucose tolerance (NGT) at Week 48 OR change from IGT at baseline to NGT at Week 48. CFRD: 2-hour post-OGTT blood glucose level ≥200 mg/dL or fasting blood glucose level ≥126 mg/dL; IGT: 2-hour post-OGTT blood glucose level ≥140 to <200 mg/dL and fasting blood glucose level <126 mg/dL; NGT: 2 hour post-OGTT blood glucose level <140 mg/dL and fasting blood glucose level <126 mg/dL.
Time Frame: Baseline, Week 48
Population: FAS. Here, "Overall Number of Participants Analyzed" signifies the number participants with non-missing dysglycemia categorization at Week 48 among participants with abnormal glucose tolerance at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 53
percentage of participants | 37.7 [24.8 to 52.1]

3. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 52
Population: Safety set included all participants who received at least 1 dose of study drug in the treatment period.
Measure: Count of Participants; unit: Participants
Groups:
- ELX/TEZ/IVA: Participants received ELX 200 mg/TEZ 100 mg/IVA 150 mg in the morning and IVA 150 mg in the evening.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 69
Participants
  Participants with TEAEs | 67
  Participants with SAEs | 6

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 52
Arm/Group | ELX/TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/69
Serious Adverse Events (participants affected / at risk) | 6/69
Other Adverse Events (participants affected / at risk) | 62/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ELX/TEZ/IVA (N=69)
Gastritis (Gastrointestinal disorders) | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ELX/TEZ/IVA (N=69)
Abdominal pain (Gastrointestinal disorders) | 9
Abdominal pain upper (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 5
Pyrexia (General disorders) | 16
Immunisation reaction (Immune system disorders) | 6
COVID-19 (Infections and infestations) | 22
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 10
Influenza (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 15
Rhinitis (Infections and infestations) | 7
Tonsillitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 7
Blood creatine phosphokinase increased (Investigations) | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 4
Headache (Nervous system disorders) | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 12
Acne (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT04599465/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT04599465/SAP_001.pdf